CLINICAL TRIAL: NCT02872194
Title: Evaluation of the Stinging Potential of Products in Human Eyes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: 17913
Record Dates: First submitted 2016-08-03; First posted 2016-08-19 (Estimated); Last update posted 2018-12-12 (Actual); Status verified 2018-12

CONDITIONS: Sunscreen Agents

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Suncare agent A + control (Experimental): Application of control and test product into one of the subjects two eyes.
  Interventions: Drug: BAY987516, Y55-170; Drug: Standard shampoo mixture (control)
- Suncare agent B + control (Experimental): Application of control and test product into one of the subjects two eyes.
  Interventions: Drug: BAY987516, X72-151; Drug: Standard shampoo mixture (control)
- Suncare agent C + control (Experimental): Application of control and test product into one of the subjects two eyes.
  Interventions: Drug: BAY987516, Y49-034; Drug: Standard shampoo mixture (control)

INTERVENTIONS:
Drug: BAY987516, Y55-170 — 10 uL in one eye
  Arms: Suncare agent A + control
Drug: BAY987516, X72-151 — 10 uL in one eye
  Arms: Suncare agent B + control
Drug: BAY987516, Y49-034 — 10 uL in one eye
  Arms: Suncare agent C + control
Drug: Standard shampoo mixture (control) — 10 uL in one eye

SUMMARY:
The objective of this study was to compare the human eye stinging potential of experimental formulas and an industry standard shampoo mixture. The study was conducted under the supervision of a Board Certified Ophthalmologist. The study design was a three cell, single blind study. Subjects were given the industry standard shampoo mixture in one eye and an exploratory sunscreen in the other as according to the randomization schedule.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects, aged 18 to 65 years
* No medical conditions of the eyes as determined by the subjects' medical history and confirmed by ophthalmologist
* Subjects do not wear contact lenses or, if he/she does wear contact lenses, is willing to refrain from wearing these during the day of and day after the study
* Subject is willing to have the test materials instilled into the eyes and follow all protocol requirements
* Subject is willing to refrain from using false eyelashes of any type or any topical prescription, OTC or cosmetic products on their eyes, eyelids, eyelashes or the peri-orbital areas of the face on the day of the study.
* Subjects should refrain from use of make-up on testing day

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2014-09-05 (Actual); Primary Completion 2014-09-06 (Actual); Study Completion 2014-09-06 (Actual)

PRIMARY OUTCOMES:
Subjective discomfort in the eye was assessed based on questions by an Ophthalmologist to the subject using a 5-category intensity scale | up to 24 hours after instillation
Tearing/Lacrimation was assessed by the Ophthalmologist using a 5-category assessment score | up to 24 hours after instillation
Objective inflammation was assessed by the Ophthalmologist using a 5-category assessment score | up to 24 hours after instillation
Post installation eye effects were assessed using a 5-category intensity score | up to 24 hours after instillation

SECONDARY OUTCOMES:
Number of adverse events as a measure of safety and tolerability | at 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- St. Petersburg, Florida, United States

REFERENCES:
- See also: Related Info — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_BSP_7261&studyid=2860&filename=17913_Study%20Synopsis_CTP.pdf